CLINICAL TRIAL: NCT05854576
Title: Markers of Metabolism and Vascular Acess Outcomes in ESRD in[Single Centre Study]
Brief Title: Markers of Metabolism and Vascular Access in ESRD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soad Elsayed Abu douh (Other)
Responsible Party: Sponsor-Investigator, Soad Elsayed Abu douh, asoad381@gmail.com, Assiut University
Organization: Assiut University (Other)
Other Study IDs: mineral metabolism in ESRD
Record Dates: First submitted 2023-04-08; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Disorders of Calcium and Bone Metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vascular acess — AVF

SUMMARY:
Aim of the study is to determine the association of markers of mineral metabolism with vascular access out come (maturation, patency of vascular access[AVF,AVG])To verify the relationship between vascular access complication (AVF,AVG) and lower levels of 25(OH)D, higher levels of fibroblast growth factor 23 (FGF23) and serum calcium, phosphorus, parathyroid hormone (PTH) in patients with ESRD on regular hemodialysis.

DETAILED DESCRIPTION:
Maintaining patent vascular access is essential for patients with end-stage renal disease (ESRD) on hemodialysis (HD) to prevent life-threatening technique failure. Access complications result in a high burden of hospital admissions, procedures, and costs for patients on HD.

, The pathophysiologic mechanisms underlying vascular access complications are poorly understood. Discovery of potential predictors and subsequent targets for intervention could help design new preventive strategies.Abnormalities in mineral homeostasis are common in patients with ESRD and are associated with numerous adverse outcomes including vascular calcification, inflammation, and mortality.

The Klotho gene encodes for a transmembrane protein, acting as a co-receptor for fibroblast growth factor-23 (FGF23) . The main functions of FGF23 signaling in the kidney are the suppression of vitamin D hormone synthesis, and the suppression of renal tubular phosphate reabsorption .

Impaired excretion of phosphorus due to low kidney function raises fibroblast growth factor 23 (FGF23). FGF23 decreases conversion of 25-hydroxy vitamin D (25(OH)D) to its active 1,25D form, causing calcium to fall and parathyroid hormone(PTH) to rise The development of secondary hyperparathyroidism lead to increased calcium and phosphate release from bones to the blood, causing the deposition of calcium and phosphate in the intima-media layer of arterial wall. and eventuating vascular calcification in these patients. the calcifications might be encountered in the upper extremity arteries in cases with ESRD .Thus, a decrease in the quality of fistula occurs in these tracts utilized frequently at the arteriovenous fistula (AVF) operations. Thes complex interplay of factors may promote vascular disease through multiple pathways including calcification, endothelial dysfunction, inflammation, activation of the renin-angiotensin-aldosterone system and others are involved. Deficiency of 25(OH)D among patients with ESRD is above 80%.1,25D or its analogs are frequently administered to patients with ESRD to overcome the adverse effects. low 25(OH)D associates with mortality in HD patients.

Vitamin D deficiency has been associated with hypertension, insulin resistance, viral and bacterial infection risk, and multiple organ damage due to systemic inflammation.

Despite consistent associations of disordered mineral homeostasis and vascular outcomes in ESRD, few studies have investigated the role of these factors in vascular access out comes

ELIGIBILITY:
Inclusion Criteria:

1. patient above the age of 18years old.
2. patient on regular hemodialysis with vascular access(AVF,AVG)
3. patient with Abnormalities in mineral metabolisms.
4. Patient secondary, Tertiary hyperparathyroidism.

Exclusion Criteria:

1. patient <18 years old
2. patient with primary hyperparathyroidism

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Despite consistent associations of disordered mineral homeostasis and vascular outcomes in ESRD, few studies have investigated the role of these factors in vascular access outcomes.
  Thes complex interplay of factors may promote vascular disease through multiple pathways including calcification, endothelial dysfunction, inflammation, activation of the renin-angiotensin-aldosterone system and others are involved(15-16),
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
association of markers of mineral metabolism with vascular access out come[maturation and patency of vascular access[AVF,AVG]] .To verify the relationship between vascular access complication (AVF,AVG) | baseline
  Aim of the study is to determine the association of markers of mineral metabolism with vascular access out come[maturation, and patency] .To verify the relationship between vascular access complication (AVF,AVG) and lower levels of 25(OH)D, higher levels of fibroblast growth factor 23 (FGF23) and serum calcium, phosphorus, parathyroid hormone (PTH) in patients with ESRD on regular hemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eman mohammed, Principal Investigator — Assiut University

REFERENCES:
- [Background] Gardezi AI, Karim MS, Rosenberg JE, Scialla JJ, Banerjee T, Powe NR, Shafi T, Parekh RS, Yevzlin AS, Astor BC. Markers of mineral metabolism and vascular access complications: The Choices for Healthy Outcomes in Caring for ESRD (CHOICE) study. Hemodial Int. 2020 Jan;24(1):43-51. doi: 10.1111/hdi.12798. Epub 2019 Dec 1. PMID 31789482